CLINICAL TRIAL: NCT01393223
Title: A Single-Center, Double-Blind, Randomized, Dose-Ranging, Placebo Controlled Trial Comparing the Safety, Tolerability and Efficacy of LP-08 With Placebo in Subjects With Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS)
Brief Title: Evaluation of Intravesical LP08 in Patients With Interstitial Cystitis/Painful Bladder Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lipella Pharmaceuticals, Inc. (Industry)
Collaborators: Corewell Health East (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PhaseII LP-08 IC/BPS
Record Dates: First submitted 2011-07-07; First posted 2011-07-13 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Interstitial Cystitis
Keywords: Interstitial Cystitis; Painful Bladder Syndrome; Bladder Pain Syndrome; Liposome; LP-08
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LP-08 80mg (Active Comparator): 4 weekly intravesical administration of LP-08 80mg
  Interventions: Drug: LP-08 80mg
- LP-08 20mg (Active Comparator): 4 weekly intravesical administration of LP-08 20mg
  Interventions: Drug: LP-08 20mg
- Normal Saline (Placebo Comparator): Four weekly normal saline intravesical administration
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: LP-08 80mg — Intravesical instillation of 80mg LP08
  Arms: LP-08 80mg
Drug: Normal saline — Intravesical instillation of normal saline
  Arms: Normal Saline
Drug: LP-08 20mg — Intravesical instillation of 20mg LP08
  Arms: LP-08 20mg

SUMMARY:
The purpose of this study is to assess the safety and tolerability of two doses of LP08 compared to placebo. Hypothesis: Safety of the LP-08 therapy will not be significantly different from the placebo group. Secondary Efficacy Endpoints: A matched-pair data analysis design will be employed, i.e. the measured outcomes will be subjects' improvements in quantitative and qualitative measures of the disease condition being assessed prior to and after LP-08 instillations at four and eight weeks follow-up visits

DETAILED DESCRIPTION:
This is a single-center, dose-ranging, placebo-controlled, double-blind, randomized study including male and female subjects with interstitial cystitis/bladder pain syndrome (IC/BPS) as determined by a physician using the current diagnostic criteria for IC/BPS. A total of 36 subjects will be enrolled at up to five (5) study sites in the U.S. Enrollment is expected to be completed within one year of initiating the study. The study is comprised of two parts. The first part of the study is a dose-ranging, randomized, double-blind, placebo-controlled study evaluating the safety, tolerability and efficacy of LP-08 at 20 mg and 80 mg doses as compared with placebo. The second part of the study is an Open Label Extension study of the safety, tolerability and efficacy of LP-08 80 mg. Subjects randomized to the placebo control group must have completed the randomized portion study, including the eight week follow-up period, to be eligible for the Open Label Extension.

ELIGIBILITY:
Inclusion Criteria:

A patient is deemed suitable for inclusion in the study if the patient meets the following criteria:

1. Male or female at least 18 years of age
2. IC/BPS diagnosed by a health care provider based the following criteria:

   Complaint of suprapubic pain related to bladder filling, accompanied by other symptoms such as increased daytime and night time frequency, in the absence of proven urinary infection or other obvious pathology Have had IC/BPS symptoms for at least six months Score of ≥ 12 on the ICSI/PI at baseline Urinary frequency > 10 times a day by self-report and confirmed on baseline three-day voiding diary Have IC/BPS that in the judgment of the investigator has been stable in the previous 30 days IC/BPS-related pain defined as a score of > 3 cm and < 9 cm on the pain VAS where 0 is no pain and 10 is maximum pain
3. Have had inadequate clinical responses with conservative treatments, which may include one or more of the following: 1) timed voiding and behavioral modification therapy, 2) dietary restrictions, 3) stress reduction and/or 5) oral therapy with any of the following medications:

   Antidepressants Antihistamines Antimuscarinic and anticholinergic agents Alpha adrenergic blockers Analgesics Pentosan polysulfate
4. Women of childbearing potential: have a negative urine pregnancy test at screening, and must agree to use an acceptable from of contraception (oral contraceptives, intrauterine or double barrier methods), as agreed to by the investigator, during the study period
5. Provide signed informed consent
6. Subject agrees to be available for the follow-up evaluations as required by the protocol

Exclusion Criteria:

Patients are excluded from enrollment in the study if any of the following are true:

1. Currently pregnant or breastfeeding, or plan to become pregnant during the course of the study
2. Have received investigational products or devices within 30 days prior to screening visit
3. Have received intravesical therapy or bladder hydrodistention within 30 days prior to screening visit. Intravesical instillations may include liquid or drug delivery devices, pentosan polysulfate sodium, lidocaine, steroid, heparin, chondroitin and any combination or additional formulation.
4. Have participated in IC/BPS research trial within 90 days prior to screening visit or has not returned to baseline if participated in IC/BPS research trial greater than 90 days prior to screening visit
5. Have received any of the following medication within 30 days of screening visit, unless such medications have been administered at a stable dose during this month and are expected to remain at a stable dose throughout the study:

   Antidepressants Antihistamines (use of antihistamines as needed for allergies is allowed) Anticonvulsants Antimuscarinic and anticholinergic agents Alpha adrenergic blockers Pentosan polysulfate sodium Oral chondroitin
6. Have indicated use of > 70 mg of morphine equivalents of opioids per week to control their IC/BPS pain within 30 days prior to screening, or are expected to require this level of IC/BPS pain control during the study period
7. Previous augmentation cystoplasty, cystectomy, neurectomy (i.e., hypogastric nerve plexus ablation). Bladder botulinum toxin injections within nine months prior to screening.
8. Sacral and/or pudendal nerve neuromodulation device (Interstim) within the last 6 months. Subjects would not be excluded if they had Interstim greater than 6 months ago and is on a stable setting within the past 90 days
9. Percutaneous Tibial Nerve Stimulation (PTNS) treatment within the past 90 days
10. Evidence of renal impairment (creatinine > two times the upper limit of normal at Visit 1), hepatic impairment (AST or ALT > three times the upper limit of normal at Visit 1), clinically significant cardiovascular, respiratory, or psychiatric diseases per investigator's judgment
11. Post-void residual (PVR) urine volume of > 150 mL at screening
12. Any condition that in the judgment of the investigator would interfere with the patient's ability to provide informed consent, comply with study instructions, place the patient at increased risk, or which might confound the interpretation of the study results
13. Previously received intravesical liposomes
14. Urinary tract or prostatic infection in the past 90 days before study entry
15. Active genital herpes or vaginitis
16. Urethral diverticulum
17. Pelvic malignancy within the past five years
18. History of cyclophosphamide or chemical cystitis, or tuberculosis or pelvic radiation
19. History of bladder or prostate tumors (benign or malignant)
20. Uncontrolled diabetes
21. Has any condition that would preclude treatment due to contraindications and/or warnings in the product labeling

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-14 (Actual)

PRIMARY OUTCOMES:
Safety of Intravesical LP08: number/severity of adverse events | Up to 31 weeks following treatment
  The number/severity of adverse events throughout the study

SECONDARY OUTCOMES:
Efficacy Voids Per Day (VPD) | 2, 4, 8, 16, 24 weeks following treatment
  The change in voids per day (urinary frequency) as measured on a 3 day voiding diary
Efficacy Global Response Assessment (GRA) | 4, 8, 16, 24 weeks following treatment
  Reporting a "moderate" or "marked" improvement on the GRA
Efficacy Symptom | 2, 4, 8, 16, 24 weeks following treatment
  The change in the symptoms and problems of interstitial cystitis from the baseline as measured by the O'Leary-Sant Interstitial Cystitis Symptom Index
Efficacy Visual Analog Scale (VAS) | 2, 4, 8, 16, 24 weeks following treatment
  The change in pain as recorded on the VAS
Efficacy Diary | 2, 4, 8, 16, 24 weeks following treatment
  The change from baseline in average voided volume, urgency and nocturia episodes per day as measured on a 3 day voiding diary

CONTACTS AND LOCATIONS:
Locations (1):
- William Beaumont Hospitals, Royal Oak, Michigan, United States